CLINICAL TRIAL: NCT03598569
Title: Dyspnea Evaluated by a Qualified Examiner in Patients With Lung Diseases
Brief Title: Auto-evaluation of Dyspnea
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: Autodyspnea
Record Dates: First submitted 2018-07-15; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-06

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- lung cancer
  Interventions: Other: dyspnea
- other lung diseases
  Interventions: Other: dyspnea

INTERVENTIONS:
Other: dyspnea — dyspnea assessment
  Other Names: evaluation

SUMMARY:
The primary aim of this study was to compare patients-rated evaluation and caregiver's assessment of dyspnea with the standard tools in pulmonology unit (Borg scale and visual analog scale) and the secondary aim was to performed an analysis depending on the diseases (lung cancer vs. other lung diseases) and to verify the agreement between the evaluation between both visual analog scale and modified Borg scale.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 and
* to have a diagnosis of acute or chronic respiratory disease

Exclusion Criteria:

* mental or cognitive disorders
* inability to understand the local language

Age Groups: Child, Adult, Older Adult
Study Population: all lung diseases
Sampling Method: Non-Probability Sample
Enrollment: 271 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
visual analog scale | 3 seconds
borg scale | 3 seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No